CLINICAL TRIAL: NCT01332708
Title: Cholinergic Status and the Metabolic Syndrome
Acronym: Choliner stat
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Prof Berliner Shlomo, Tel-Aviv Sourasky Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TASMC-11-SB-10-538-CTIL
Record Dates: First submitted 2011-04-07; First posted 2011-04-11 (Estimated); Last update posted 2011-04-11 (Estimated); Status verified 2011-04

CONDITIONS: Overweight; Obese
Keywords: high complex carbohydrates; hypocaloric diet; cholinergic status; overweight; obese
MeSH Terms: conditions — Overweight; Obesity

ARMS (1):
- Obese and overweight subjects (Experimental): The participants are overweight and obese people with and without metabolic syndrome that will participate in diet groups.
  Interventions: Behavioral: high complex carbohydrates diet given in a diet group

INTERVENTIONS:
Behavioral: high complex carbohydrates diet given in a diet group — diet groups that meet every week for eight weeks or more.

SUMMARY:
The investigators aims in the current study are to examine whether the cholinergic status should be considered as another risk factor for the metabolic syndrome and it's co-morbidities and to test the effect of a hypocaloric high complex carbohydrates diet on the cholinergic status of overweight and obese adults with and without the metabolic syndrome.

DETAILED DESCRIPTION:
Intervention studies have demonstrated that the autonomic disturbances of the metabolic syndrome may be reversible. A reduction in body weight induced by a hypocaloric diet exerts a marked reduction in sympathetic activity in obese people with or without metabolic syndrome. Incorporation of regular, moderate intensity aerobic exercise training during a dietary weight loss program does not confer additional benefits on resting sympathetic neural activity, compared with weight loss by diet alone. A new method has been developed to examine the sympathetic-parasympathetic status of an individual - the cholinergic status. Cholinergic Status represents the total soluble circulation capacity for acetylcholine hydrolysis. Higher cholinergic status means the individual is more sympathetic .

A cross sectional study that took place in Tel Aviv Sorasky medical center and included 632 participants found that the cholinergic status is related to metabolic syndrome parameters in a dose response manner and that it correlates significantly with glucose,HbA1c, lipid profile and hs-CRP.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 25kg/m2
* Stable weight (±1kg)in the previous six months
* Non smokers

Exclusion Criteria:

* Type II diabetes
* Hypertension pharmacologically treated
* Cardiovascular disease
* Renal disease
* Cirrhosis and end-stage liver failure
* Thyroid disease
* Cerebrovascular disease
* Cancer
* Autoimmune disease
* Chronic inflammatory disease
* Surgery or heart catheterization in the previous six months
* Use of drugs known to affect measured parameters

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-04; Primary Completion 2011-08 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
total soluble circulation capacity for acetylcholine hydrolysis | 8 weeks or more

SECONDARY OUTCOMES:
Inflammatory markers | 8 weeks or more
  hs-CRP, ESR, Fibrinogen, IL-1b, IL-6, TNF-α
ROTEM - rotation thromboelastometry | 8 weeks or more
  ROTEM documents the interaction of platelets with the coagulation factors from initial platelet-fibrin interaction, through platelet aggregation, clot strengthening and fibrin cross-linking to eventual clot lysis. Within 30 min, a ROTEM tracing provides information on clotting factor activity, platelet function and any clinically significant fibrinolysis.
Metabolic markers | 8 weeks or more
  Fasting Glucose, HbA1c,Insulin, lipid profile